CLINICAL TRIAL: NCT07304427
Title: A Prospective, Multicenter, Post-market Clinical Investigation to Evaluate the Pre-dilation Safety and Effectiveness of Alwide Plus Balloon Catheter of MicroPort CardioFlow in Transcatheter Aortic Valve Replacement
Brief Title: Alwide Plus China Post-market Clinical Investigation
Status: Completed | Type: Observational
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Alwide Plus-2024
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Severe Aortic Stenosis; Transcatheter Aortic Valve Replacemen
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alwide Plus: Paitents perfomed TAVR and have Alwlide Plus Balloon Catheter pre-dilaton or post-dilation

SUMMARY:
This is a prospective, single-arm, multi-center, post-market registry study conducted in China. The purpose is to evaluate the safety and effectiveness of the AlwideTM Plus balloon catheter for pre-dilatation of the aortic valve during TAVR in the real-world setting.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety and effectiveness of the Alwide Plus balloon catheter for pre-dilatation of the aortic valve during in transcatheter aortic valve replacement in the real-world setting, with TAVI device success at immediate post-procedure as the primary endpoint. The immediate post-procedural pre-dilation success, all-cause mortality, stroke, bleeding, acute kidney injury, permanent pacemaker implantation, major vascular complication, valve function at post-procedure and discharge, and post-dilation success will be used as secondary endpoints.This is a prospective, multi-center, post market clinical investigation. 75 patients will be enrolled in this clinical investigation. All subjects will undergo telephone follow-up at 30 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Severe aortic stenosis verified by echocardiogram: mean transvalvular gradient≥40mmHg (1mmHg=0.133kPa), or peak aortic jet velocity≥4m/s, or aortic valve area (AVA) ≤ 1.0cm2 (or AVA index≤ 0.6cm2/m2);
* Patients, who can understand the clinical investigation purpose, voluntary agree and sign the informed consent form, and willing to comply with relevant trial assessments and clinical follow up

Exclusion Criteria:

* Aortic valve anatomy or lesion unsuitable or not necessary for balloon pre-dilation during the TAVR procedure
* TAVR procedure in trans-apical access
* Pre-implanted mechanical or bioprosthetic valve at the aortic valve position
* Acute myocardial infarction (MI) occurred in the last 30 days before the treatment；
* LVOT obstruction;
* Serious left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20%
* Echocardiographic evidence of intracardiac mass, thrombus or neoplasm；
* Unable to receive anticoagulation or antiplatelet therapy；
* Allergy to nitinol or sensitive contrast media；
* Active bacterial endocarditis or other active infection may affect the procedure；
* Aortic valve anatomy , lesion, or other situation unsuitable for the prosthesis valve implantation as assessed by the investigator team；
* Life expectancy > 12 months；
* vulnerable individuals who are unable to give informed consent/ unable to fully understand all aspects of the investigation or Severe incapacitating Alzheimer's disease；
* Patients who participated in other clinic trials of drugs or medical device before being enrolled for which the primary endpoint follow up duration has not been reached；
* Investigators determined that patients have poor compliance and can't complete the study as required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering severe aortic stenosis and requiring pre-dilation during TAVR
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with TAVI device success at immediate post-procedure | Immediate post-procedure
  TAVI device success, defined as (meeting all the following criteria):
  Freedom from mortality; Successful access, delivery, deployment, implantation of the valve, and retrieval of the delivery system; Correct positioning of the prosthetic heart valve into the proper anatomical location; Intended performance of the valves (mean gradient <20mmHg, or peak velocity <3 m/s, and no severe aortic regurgitation or paravalvular leakage).

SECONDARY OUTCOMES:
Percentage of patients with balloon pre-dilation success | Immediate post-procedure
  defined as successful access, delivery and dilation the aortic valve, and retrieval for the AlwideTM Plus balloon catheter
Percentage of paitents with balloon post-dilation success | Immediate post-procedure
  defined as successful access, delivery and dilation the transcatheter aortic valve, and retrieval for the AlwideTM Plus balloon catheter
Incidence of all-cause mortality, disabling and non-disabling stroke, life-threatening or disabling bleeding, major bleeding, acute kidney injury(AKIN≥2), major vascular complications and new permanent pacemaker implantation | Immediate post-procedure and 30 days post-procedure
  Definition following VARC-2 criteria
Prosthetic valve performance-mean transvalular pressure gradient | Immediate post-procedure and discharge(within 7 days post-procedure)
  Prosthetic valve performance-mean pressure gradient(assessed by echocardiography), unit -mmHg
Prosthetic valve performance-orifice area | Immediate post-procedure and discharge(within 7 days post-procedure)
  Prosthetic valve performance-orifice area(assessed by echocardiography), unit -cm2
Prosthetic valve performance-valve regurgitation(intra- and para valvular leakage) | Immediate post-procedure and discharge(within 7 days post-procedure)
  Prosthetic valve performance-valve regurgitation(intra- and para valvular leakage), none/trace/mild/moderate/severe

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Guangdong Provincial People's Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No